CLINICAL TRIAL: NCT02460250
Title: Evaluation of Liver Grafts With FibroScan® Before Organ Retrieval in Patients With Brain Death
Acronym: FIBROSCAME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: I12033 FIBROSCAME
Record Dates: First submitted 2015-05-13; First posted 2015-06-02 (Estimated); Last update posted 2019-10-24 (Actual); Status verified 2019-10

CONDITIONS: Tissue and Organ Harvesting; Liver Transplantation; Brain Death
Keywords: Tissue and Organ Harvesting; Liver graft; Brain Death; FibroScan®
MeSH Terms: conditions — Brain Death

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fibroscan (Experimental): All included patients will undergo a Fibroscan (either Fibroscan Touch model or 402 model which enable CAPTM data extraction) once all eligibility criteria have been checked. Liver recipients will be followed up during one year. Biological and medical data used by all transplant sites for the follow-up of transplant patient will be collected
  Interventions: Procedure: Fibroscan

INTERVENTIONS:
Procedure: Fibroscan — All included patients will undergo a Fibroscan (either Fibroscan Touch model or 402 model which enable CAPTM data extraction) once all eligibility criteria have been checked.

SUMMARY:
According to the French Biomedicine Agency annual report on retrieval activities and transplants, 1,164 liver transplants were performed in 2011 and 1,161 in 2012. If the amount of brain death donors and retrieved liver grafts appears relatively stable, it remains clearly insufficient compared to the increasing number of patients on the waiting list for liver transplantation (2,462 in 2011). The median time on the waiting list before liver transplantation which was established from the cohort of patients registered between 2007 and 2011 (excluding patients registered for emergency transplantation and for living related-donor transplantation) increased significantly from 4.4 months between 2007 and 2009 to 6.6 months between 2010 and 2011. In order to compensate for the lack of liver grafts, donors acceptance criteria were broadened. For example, alternative transplantation lists were created with liver grafts coming from so-called "marginal" donors. However, despite these efforts, livers were retrieved on only two out of three brain death donors, i.e. in 1,572 and 1,589 organ donors in 2011 and 2012, respectively. This is unfortunately not enough to meet the increasing needs in liver grafts and a growing number of patients wait each year for transplant. Strategic lines of improvement were defined in order to meet the "2012-2016 transplant perspective" which targets 5,700 transplants carried out in 2015 (+5% every year, all transplants included, with 5,023 transplants in 2012).

According to the last consensus conference on liver transplantation of the HAS (French High Authority of Health) the assessment of the degree of macrovacuolar and microvacuolar steatosis determines the possibility to retrieve the graft or not. Liver steatosis consists in an accumulation of fatty droplets in hepatocytes. Its prevalence is high, ranging from 16% to 31% in the general population, and increases up to 46% in heavy drinkers and to 50-80% in the obese population. Steatosis results mostly from alcohol consumption and from metabolic syndrome (obesity, type 2 diabetes, hypertriglyceridemia) called non-alcoholic fatty liver disease (NAFLD), and is more rarely secondary to viral hepatitis or exposure to certain medications. NAFLD involves up to 30% of the population in Western countries and its prevalence is increasing. NAFLD may lead to asymptomatic steatosis, but also to steatohepatitis or advanced fibrosis including cirrhosis and its complications Accordingly, the improvement of liver grafts selection based on objective quantitative criteria which takes into account the degree of liver steatosis appears crucial to increase the number of hepatic transplants.

DETAILED DESCRIPTION:
Medical procedure: Fibroscan® based on vibration control transient elastography (VCTETM) with evaluation of controlled attenuation parameter (CAP™) by ultrasounds (Echosens, Paris, France).

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years with recognized clinical brain death confirmed by clinical examination, who are considered for organ retrieval and clinically stable to achieve the retrieval procedure

Exclusion Criteria:

* Personal objection to organ retrieval and clinical research expressed during lifetime and registered in the Registre National des Refus (French registration of all refusals to organ donation)
* Family objection to liver retrieval after donor's death
* Ongoing pregnancy when brain death is declared
* For FT and ST measurements included in the panel FibroMaxTM, 4 exclusion criteria are defined specifically (Acute hepatitis or cytolysis with ALT higher than 622 IU/L, acute or chronic hemolysis, extrahepatic cholestasis, sepsis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 740 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2017-11-09 (Actual); Study Completion 2018-11-09 (Actual)

PRIMARY OUTCOMES:
Controlled Attenuation Parameter™ (CAP™) measurement | 1 Day
  Evaluation of the diagnostic accuracy of the CAP™ measured with Fibroscan® to objectively reflect the degree of liver steatosis, a parameter which can be used as an aid in selecting liver grafts before retrieval in donors with brain death (DBD).

SECONDARY OUTCOMES:
Liver Stiffness (LS) measurement | 1 Day
  Evaluation of the diagnostic accuracy of LS measured with Fibroscan® to objectively reflect the degree of fibrosis and steatosis, a parameter which can be used as an aid in selecting liver grafts before retrieval in DBD
Controlled Attenuation Parameter™ (CAP™) measurement | 1 week
  Determination of the prognostic value of CAP™ in terms of survival of liver grafts at one week after transplantation
Liver Stiffness (LS) measurement | 1 week
  Determination of the prognostic value of LS in terms of survival of liver grafts at one week after transplantation
Liver Stiffness (LS) measurement | 1 month
  Determination of the prognostic value of LS in terms of survival of liver grafts at one month after transplantation
Controlled Attenuation Parameter™ (CAP™) measurement | 1 month
  Determination of the prognostic value of CAP™ in terms of survival of liver grafts at one month after transplantation
Liver Stiffness (LS) measurement | 1 year
  Determination of the prognostic value of LS in terms of survival of liver grafts at one week, one month and one year after transplantation
Controlled Attenuation Parameter™ (CAP™) measurement | 1 year
  Determination of the prognostic value of CAP™ in terms of survival of liver grafts at one week, one month and one year after transplantation
Fibrosis measurement | 1 Day
  evaluate the diagnostic a accuracy of FibroTest in selecting liver grafts before retrieval in DBD by comparing with 1) histological data obtained with liver biopsy (degree of steatosis, degree of fibrosis) and with 2) CAPTM/LS
Steatosis measurement | 1 Day
  evaluate the diagnostic a accuracy of SteatoTest in selecting liver grafts before retrieval in DBD by comparing with 1) histological data obtained with liver biopsy (degree of steatosis, degree of fibrosis) and with 2) CAPTM/LS
Fibrosis measurement | 1 month
  Determination of the short-term prognostic values of FibroTest in terms of survival of liver grafts at one month after transplantation
Steatosis measurement | 1 month
  Determination of the short-term prognostic values of SteatoTest in terms of survival of liver grafts at one month after transplantation
Fibrosis measurement | 1 year
  Determination of the short-term prognostic values of FibroTest in terms of survival of liver grafts at one year after transplantation
Steatosis measurement | 1 year
  Determination of the short-term prognostic values of SteatoTest in terms of survival of liver grafts at one year after transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas PICHON, MD, Principal Investigator — University Hospital, Limoges
Locations (19):
- France (19):
  - University Hospital, Amiens
  - University Hospital, Angers
  - University Hospital, Besançon
  - University Hospital, Bordeaux
  - University Hospital, Brest
  - University Hospital, Caen
  - Estaing University Hospital, Clermont-Ferrand
  - AP-HP Henri MONDOR, Créteil
  - University Hospital, Grenoble
  - University Hospital, Lille
  - University Hospital, Limoges
  - Croix Rousse Hospital, Lyon
  - Nice University Hospital, Nice
  - AP-HP Kremlin Bicêtre, Paris
  - University Hospital, Poitiers
  - Univesity Hospital, Reims
  - University Hospital, Rennes
  - University Hospital, Tours
  - University Hospital, Vandœuvre-lès-Nancy